CLINICAL TRIAL: NCT06613282
Title: A Randomized Single-blind Study of LI-TMS and AVS for Stroke Recovery in Healthy Participants with the Evaluation of the Effect on the Subject Using EEG and the Following Testing.
Brief Title: A Randomized, Single-blind Trial of LI-TMS and AVS for Stoke Recovery in Healthy Participants (Phase 1).
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Siberian Scientific Research and Test Center for Biomedical Engineering (Other)
Collaborators: Novosibirsk State Medical University (Other)
Responsible Party: Principal Investigator, Viktor Anatolyevich Drobyshev, Doctor of Medical Sciences, Professor of the Department of Hospital Therapy and Medical Rehabilitation at the Novosibirsk State Medical University, Head of the Physiotherapy Department at City Clinical Hospital No. 2, Siberian Scientific Research and Test Center for Biomedical Engineering
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LI-TMS and AVS for recovery
Record Dates: First submitted 2024-09-17; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Recovery Methods; Rehabilitation Program; Stroke, Ischemic; Stroke
Keywords: Low Intensity Transcranial Magnetic Stimulation; audio-visual stimulation; AVS; recovery after stroke; stroke rehabilitation; LI-TMS
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Photic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LI-TMS and AVS (Experimental): Participants receive low-intensity transcranial magnetic stimulation interventions with audio-visual stimulation for 14 days. On days 6, 7, 13, and 14 of the study, participants will not receive any interventions. Participants will be screened and tested on days 1 and 14 of treatment and two weeks after the end of the intervention.
  Interventions: Device: Low Intensity Transcranial Magnetic Stimulation; Device: Auditory and visual stimulation
- Control (No Intervention): Participants receive no interventions for 14 days. Participants will be screened and tested on days 1, 14 and 28.

INTERVENTIONS:
Device: Low Intensity Transcranial Magnetic Stimulation — * Magnetic stimulation frequency range: 0.1 - 700 Hz.
  * Amplitude of the magnetic field at a short distance from the magnetic coil: 1-5 milliTesla.
  * Emitter coil dimensions: ⌀28×26 mm.
  * Number of emitter coils: 32 coils.
  * Covering the entire scalp of a human head with 32 coil emitters.
  Other Names: LI-TMS
  Arms: LI-TMS and AVS
Device: Auditory and visual stimulation — * Frequency range of light stimulation: 0.1 - 60 Hz.
  * Audio stimulation frequency range: 20 - 2000 Hz.
  * Sound level: 70 Decibel.
  * The wavelength range of visual stimulation: red - 620 - 760 nm; green - 510 - 550 nm; blue - 450 - 480 nm.
  * Illuminance: 300 - 350 lx.
  Arms: LI-TMS and AVS

SUMMARY:
This randomized, controlled, single-blind clinical pilot study investigates the therapeutic potential of low-intensity repetitive transcranial magnetic stimulation (LI-TMS) and audio-visual stimulation (AVS) and newly offered interventional protocols in healthy participants for further research on stroke rehabilitation and therapeutic effects.

The goal of this clinical trial is to learn if the intervention can be used in the future treatment of patients recovering after stroke. It will also learn about the safety of low-intensity repetitive transcranial magnetic stimulation and audio-visual stimulation.

The main questions it aims to answer are:

Does intervention with LI-TMS and AVS influence the parameter Work Efficiency (WE) of the participant? Does intervention with LI-TMS and AVS influence the parameter Warming-up work indicator (WU) of the participant? Does intervention with LI-TMS and AVS influence the parameter Psychological Stability (PS) of the participant? Does intervention with LI-TMS and AVS influence the parameter Perceptual Accuracy (Tv) of the participant? Does intervention with LI-TMS and AVS affect changes in the participants electroencephalogram parameters? The researchers will compare the results of LI-TMS and AVS intervention to a control group that received no intervention but only underwent an examination to evaluate the effects of the interventions.

Participants will:

Receive interventions from LI-TMS and AVS every day for 2 weeks with a weekend break on Saturday and Sunday.

Attend the clinic 3 times during the trial and undergo testing and screening. The first clinic visit is before the intervention course. The second clinic visit will be the day immediately following the end of the two-week intervention course. The third visit will be two weeks after the second visit.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability worldwide, significantly impacting individuals; quality of life and their ability to perform daily activities. Rehabilitation is critical for stroke survivors as it aims to restore function, improve mobility, and enhance overall well-being.

Auditory-visual stimulation (AVS) is a stroke rehabilitation technique that combines auditory and visual stimuli to promote cognitive and motor recovery. This approach is based on the principles of neuroplasticity, which suggest that engaging multiple senses through receptor systems can promote brain plasticity and recovery after neurological injury such as stroke.

Transcranial Magnetic Stimulation (TMS) is a promising technique in stroke rehabilitation that involves applying magnetic fields to the scalp, which induces electrical currents in specific brain regions. This method is believed to facilitate neuroplasticity, the brains ability to reorganize itself by forming new neural connections.

LI-TMS is a variant of TMS that uses lower intensity magnetic fields. This technique is designed to minimize discomfort while still promoting neuroplasticity. Key aspects of LI-TMS include:

1. Safety and Tolerability: LI-TMS is generally well-tolerated, making it suitable for patients who may be sensitive to higher-intensity stimulation.
2. Potential for Long-Term Effects: Studies suggest that LI-TMS may lead to sustained improvements in motor function and cognitive abilities, even after treatment has ended.
3. Combination with Other Therapies: LI-TMS can be effectively combined with traditional rehabilitation methods, enhancing overall therapeutic outcomes.

This study aims to test the proposed interventional protocols using a prototype device for low-intensity repetitive transcranial magnetic stimulation (LI-TMS) and audio-visual stimulation (AVS) on healthy participants.

Participants in the experimental group are screened and tested upon their first visit to the hospital. Afterward, intervention courses are run five days a week for two weeks. Activities take place on Monday, Tuesday, Wednesday, Thursday and Friday while Saturday and Sunday are free. Interventions of each protocol are applied for two days in routine. At the end of the intervention course, participants are screened and tested again at the hospital and after two weeks.

The following is how the Interventional procedure goes: first, the device will be plugged in and tested, then in 5 minutes the subject sits in a comfortable chair, further a disposable hair cap is put on his/her head, a textile helmet with coil emitters is put on top of the disposable hair cap, then glasses with Red, Green, Blue Light-emitting diodes and stereo headphones. The Interventional protocol was selected in prototype software. In conformance with the selected Interventional protocol, the characteristics of the exposure signal were then set up. The button on the prototypes touch screen was pressed next. The intervention procedure was stopped when the time on the timer on the touch screen of the prototype expired. When the exposure procedure was over, the prototype was switched off and all its exposure units were taken off of the test subject in reverse order.

The study will involve two groups: an experimental group and a control group. The experimental group, consisting of 30 healthy participants, will receive a course of interventions over two weeks of days. The comparison will be made with a control group consisting of 10 healthy participants who will receive no intervention, only screening, and testing.

Interventions. Experimental: Day 1 and Day 2

1. For low-intensity transcranial magnetic stimulation, six radiating coils are placed in the temporal region above the hippocampus. A stimulation frequency of 6 Hz is applied to all emitters. The signal waveform to be used has a sinusoidal shape and bipolar type.
2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear is 440 Hz and for the right ear is 446 Hz. The signal waveform to be used has a sinusoidal shape and unipolar type.
3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye is 1 Hz and for the right eye is 7 Hz. The signal waveform to be used has a sinusoidal shape and unipolar type.
4. For colour stimulation, the left eye is exposed to blue for 6 minutes in the initial stage and green for 6 minutes in the final stage. The right eye is exposed to the colour green for 6 minutes in the initial stage and blue for 6 minutes in the final stage as well.
5. The total time duration of the procedure is 12 minutes. Experimental: Day 3 and Day 4

1. For low-intensity transcranial magnetic stimulation, six radiating coils are placed in the temporal region above the hippocampus. The frequencies of the stimulation signal are varied as follows: at the initial stage the signal frequency is 4 Hz is applied to all emitters and lasts for 6 minutes, then the frequency increases to 5 Hz for the next 6 minutes, then to 6 Hz for the next 6 minutes, then to 7 Hz for the next 6 minutes, and at the final stage the signal frequency is 8 Hz and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and bipolar type.

2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear in the initial stage is 440 Hz and for the right ear is 444 Hz, and lasts for 6 minutes. In the next stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 445 Hz, and lasts for 6 minutes. Next, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 446 Hz, and lasts 6 minutes. Then the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 447 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 448 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.

3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye in the initial stage is 1 Hz and for the right eye is 5 Hz and lasts for 6 minutes. In the next stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 6 Hz, and lasts for 6 minutes. Next, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 7 Hz, and lasts for 6 minutes. Then the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 8 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 9 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.

4. For colour stimulation, the left eye is exposed to red in the initial stage and the right eye is exposed to green, and lasts for 6 minutes. In the next stage, the left eye is exposed to the colour blue and the right eye is exposed to the colour violet and lasts for 6 minutes. Next, the left eye is exposed to the colour green and the right eye is exposed to the colour blue, and lasts for 6 minutes. Then the left eye is exposed to the colour violet and the right eye is exposed to the colour green, and lasts for 6 minutes. In the final stage, the left eye is exposed to the colour green and the right eye to the colour red, and lasts for 6 minutes.

5. The total time duration of the procedure is 30 minutes. Experimental: Day 5

1. For low-intensity transcranial magnetic stimulation, six radiating coils are placed in the temporal region above the hippocampus. Frequencies of the stimulation signal are varied as follows: in the initial stage, the carrier frequency of the signal is 8 Hz and the modulating frequency is 4 Hz, and lasts for 6 minutes. In the next stage, the carrier frequency of the signal stays 8 Hz and the modulating frequency increases to 5 Hz, and lasts for 6 minutes. Next, the carrier frequency of the signal stays 8 Hz, and the modulating frequency is increased to 6 Hz, and lasts for 6 minutes. Then the carrier frequency of the signal stays 8 Hz, and the modulating frequency is increased to 7 Hz, and lasts for 6 minutes. In the final step, the signal carrier frequency and modulating frequency are equal to 8 Hz, resulting in the signal being a regular sinusoid with a frequency of 8 Hz, and lasting 6 minutes. Carrier signal waveform - sine wave, modulating signal waveform - cosine wave. The signal type is bipolar.

2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear in the initial stage is 440 Hz and for the right ear is 444 Hz, and lasts for 6 minutes. In the next stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 445 Hz, and lasts for 6 minutes. Next, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 446 Hz, and lasts 6 minutes. Then the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 447 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 448 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.

3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye in the initial stage is 1 Hz and for the right eye is 5 Hz and lasts for 6 minutes. In the next stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 6 Hz, and lasts for 6 minutes. Next, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 7 Hz, and lasts for 6 minutes. Then the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 8 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 9 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.

4. For colour stimulation, the left eye is exposed to red in the initial stage and the right eye is exposed to green, and lasts for 6 minutes. In the next stage, the left eye is exposed to the colour blue and the right eye is exposed to the colour violet and lasts for 6 minutes. Next, the left eye is exposed to the colour green and the right eye is exposed to the colour blue, and lasts for 6 minutes. Then the left eye is exposed to the colour violet and the right eye is exposed to the colour green, and lasts for 6 minutes. In the final stage, the left eye is exposed to the colour green and the right eye to the colour red, and lasts for 6 minutes.

5. The total time duration of the procedure is 30 minutes. Experimental: Day 6 Day of no interventions. Experimental: Day 7 Day of no interventions. Experimental: Day 8

1. For low-intensity transcranial magnetic stimulation, six radiating coils are placed in the temporal region above the hippocampus. Frequencies of the stimulation signal are varied as follows: in the initial stage, the carrier frequency of the signal is 8 Hz and the modulating frequency is 4 Hz, and lasts for 6 minutes. In the next stage, the carrier frequency of the signal stays 8 Hz and the modulating frequency increases to 5 Hz, and lasts for 6 minutes. Next, the carrier frequency of the signal stays 8 Hz, and the modulating frequency is increased to 6 Hz, and lasts for 6 minutes. Then the carrier frequency of the signal stays 8 Hz, and the modulating frequency is increased to 7 Hz, and lasts for 6 minutes. In the final step, the signal carrier frequency and modulating frequency are equal to 8 Hz, resulting in the signal being a regular sinusoid with a frequency of 8 Hz, and lasting 6 minutes. Carrier signal waveform - sine wave, modulating signal waveform - cosine wave. The signal type is bipolar.
2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear in the initial stage is 440 Hz and for the right ear is 444 Hz, and lasts for 6 minutes. In the next stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 445 Hz, and lasts for 6 minutes. Next, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 446 Hz, and lasts 6 minutes. Then the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 447 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left ear stays 440 Hz and the frequency for the right ear increases to 448 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.
3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye in the initial stage is 1 Hz and for the right eye is 5 Hz and lasts for 6 minutes. In the next stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 6 Hz, and lasts for 6 minutes. Next, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 7 Hz, and lasts for 6 minutes. Then the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 8 Hz, and lasts for 6 minutes. In the final stage, the frequency for the left eye stays 1 Hz and the frequency for the right eye increases to 9 Hz, and lasts for 6 minutes. The signal waveform to be used has a sinusoidal shape and unipolar type.
4. For colour stimulation, the left eye is exposed to red in the initial stage and the right eye is exposed to green, and lasts for 6 minutes. In the next stage, the left eye is exposed to the colour blue and the right eye is exposed to the colour violet and lasts for 6 minutes. Next, the left eye is exposed to the colour green and the right eye is exposed to the colour blue, and lasts for 6 minutes. Then the left eye is exposed to the colour violet and the right eye is exposed to the colour green, and lasts for 6 minutes. In the final stage, the left eye is exposed to the colour green and the right eye to the colour red, and lasts for 6 minutes.
5. The total time duration of the procedure is 30 minutes. Experimental: Day 9 and Day 10

1. For low-intensity transcranial magnetic stimulation involved all 32 magnetic emitters located over the entire scalp area. The stimulation frequencies were as follows: the carrier signal frequency was 13 Hz, and the modulating signal frequency was determined by the operator based on the participants previously measured electroencephalogram (e.g., 9 Hz). The shape of the carrier signal was a sine wave, and the shape of the modulating signal was a cosine wave. The signal type is bipolar. Carrier signal waveform - sine wave, modulating signal waveform - cosine wave. The signal type is bipolar.

2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear is 440 Hz and for the right ear is (440 + n) Hz, where n is a frequency value determined by the operator based on the participants previously measured electroencephalogram (e.g., 9 Hz). The signal waveform to be used has a sinusoidal shape and unipolar type.

3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye is 1 Hz and for the right eye is (1 + n) Hz, where n represents a frequency value determined by the operator based on the participants previously measured electroencephalogram (e.g., 9 Hz). The signal waveform to be used has a sinusoidal shape and unipolar type.

4. For colour stimulation, the left eye is exposed to blue for 6 minutes in the initial stage and green for 6 minutes in the final stage. The right eye is exposed to the colour green for 6 minutes in the initial stage and blue for 6 minutes in the final stage as well.

5. The total time duration of the procedure is 12 minutes. Experimental: Day 11 and Day 12

1. For low-intensity transcranial magnetic stimulation involved all 32 magnetic emitters located over the entire scalp area. The stimulation frequencies were as follows: the carrier signal frequency was 25 Hz, and the modulating signal frequency was determined by the operator based on the participants previously measured electroencephalogram (e.g., 14 Hz). The shape of the carrier signal was a sine wave, and the shape of the modulating signal was a cosine wave. The signal type is bipolar. Carrier signal waveform - sine wave, modulating signal waveform - cosine wave. The signal type is bipolar.
2. For auditory stimulation, a binaural beats technique is used, where the frequency for the left ear is 440 Hz and for the right ear is (440 + n) Hz, where n is a frequency value determined by the operator based on the participants previously measured electroencephalogram (e.g., 14 Hz). The signal waveform to be used has a sinusoidal shape and unipolar type.
3. For visual stimulation, the technique of different frequencies of the signals applied to the eyes is used, where the frequency for the left eye is 1 Hz and for the right eye is (1 + n) Hz, where n represents a frequency value determined by the operator based on the participants previously measured electroencephalogram (e.g., 14 Hz). The signal waveform to be used has a sinusoidal shape and unipolar type.
4. For colour stimulation, the left eye is exposed to blue for 6 minutes in the initial stage and green for 6 minutes in the final stage. The right eye is exposed to the colour green for 6 minutes in the initial stage and blue for 6 minutes in the final stage as well.
5. The total time duration of the procedure is 12 minutes. Experimental: Day 13 Day of no interventions. Experimental: Day 14 Day of no interventions.

Control: Day 1 - Day 14 The control group does not receive any intervention for 14 days.

Participants in the experimental group and control group are screened and tested on the first day and on day fourteen and on day 28th of the study.

ELIGIBILITY:
Inclusion Criteria:

Participants must be in good general health, as verified by reviewing their medical history and physical examination. They must not have any serious illnesses that could be a barrier to the research.

Exclusion Criteria:

1. somatic and neurological diseases in the exacerbation stage;
2. presence of epileptic seizures on the EEG;
3. cognitive disorders;
4. presence of visual and hearing pathologies that prevent the sessions;
5. women during pregnancy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Work Efficiency (WE) | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  Work Efficiency (WE) is a key parameter derived from the Schulte table test that quantifies the effectiveness of a participants performance during the test. It reflects the relationship between the number of correct responses and the time taken to complete the task.
  Calculation of Work Efficiency is calculated using the following formula:
  WE= T/N.
  Where:
  N = the number of tables completed by the participant. T = Time taken to complete the test (measured in seconds). This formula indicates that Work Efficiency increases with either a higher number of correct responses or a shorter completion time.
  Measurement Units Values in the range of 30 to 50 seconds are good result. Values above 90 seconds are a negative result. Better result of WE suggest better cognitive efficiency and processing speed, while worse result may indicate difficulties in attention or visual processing.
Warming-up Work Indicator (WU) | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  Warming-up Work Indicator (WU) indicates the amount of effort or cognitive load that an individual expends during the initial phase of the test.
  Calculation of WU The WU is typically calculated based on the time taken to complete the first task of the Schulte table test compared to the overall time taken for the entire test.
  The first tasks time is compared with the average WE time. A WU ratio close to 1 indicates the best possible preparation of the participant, whereas ratios above 1 indicate that more time needs to be taken as a warm-up before optimal performance.
  WU = T1 / WE Measurement Units A result less than 1.0 is an indicator of good Warming-up Work Indicator; accordingly, the higher 1.0 this indicator is, the more the subject needs preparation for the main job.
Psychological Stability (PS) | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  Psychological Stability (PS) is a parameter derived from the Schulte table test that assesses the ability to sustain the operational activity for a long time. It reflects how well a participant can manage distractions and maintain attention throughout the test.
  Calculation:
  PS =T(n-1) /WE. Measurement Units. Psychological Stability does not have a standardized unit of measurement; rather, it is often expressed as a score or index that can be compared across individuals or populations.
  Measurement Units The result indicator less than 1.0 indicates good Psychological Stability, accordingly, the higher this indicator is, the worse the Psychological Stability of the test subject to perform the tasks.
Attention switching time (t) | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  The Test of Attention Switching Time Using Black-Red Table is a psychological assessment designed to measure the efficiency of attention switching in individuals. Attention switching time (t) refers to the duration it takes for an individual to shift their focus from one task or stimulus to another. It is a critical parameter in cognitive psychology, as it reflects the efficiency of an individuals cognitive processing and ability to manage attention in dynamic environments.
  Calculation:
  The difference between the time required to complete the last task and the sum of the time spent working on the first and the second task will be the time the subject spends switching attention from one activity to another.
  Measurement Units A shorter completion time of the Attentional Switching Time Test using the Black-Red Tables indicates better attentional switching ability.
Perceptual Accuracy (Tv) | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  The Memorize and Place Shapes task is a cognitive assessment designed to evaluate spatial memory and perceptual accuracy.
  Perceptual Accuracy (Tv) refers to the precision with which an individual can recognize and reproduce shapes after they have been memorized. This parameter is crucial in understanding cognitive functions related to memory and visual processing.
  Calculation:
  The result is an overall calculation made from the complete number of dots correctly placed on all forms. Among others, the following is calculated: Perceptual accuracy: Tv = (∑ / n) * 100, where ∑ is the total number of correctly filled-in Remember and dot test forms and n is the number of dot cards viewed. Multiply the result of the division by 100 to obtain the perceptual accuracy in percent.
  Measurement Units The higher the Perceptual Accuracy (Tv) score on the Memorise and Place Shapes test, the better the participant's visual perception.

SECONDARY OUTCOMES:
EEG | Immediately before the intervention course (at baseline), immediately after the intervention course, and 28 days after completion of the intervention course.
  Standard procedure for recording an electroencephalogram.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Drobyshev, Dr. Med. Sc., Principal Investigator — Novosibirsk State Medical University
Locations (1):
- Novosibirsk State Medical University, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underline results in a publication will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Materials will be made available 6 months after publication of the primary outcomes.
Access Criteria: Data and study materials relevant to any publication will be posted within six months of publication on this site or another open platform on the Internet which will be accessible to any interested party.